CLINICAL TRIAL: NCT06209541
Title: Tailored or Transdiagnostic ICBT with a Specific Therapist or Team Support: a Factorial Randomized Controlled Trial
Brief Title: Internet-based Cognitive Behavioral Therapy: a Factorial Randomized Controlled Trial About Treatment Content and Support
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INES
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Depression Symptoms; Anxiety Symptoms
Keywords: Internet-based cognitive behavioral therapy (ICBT); Internet intervention; Depression; Anxiety; Individually tailored; Transdiagnostic; Alliance
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: After recruitment finished, participants will be randomized to one of four groups that differ in type of treatment content (Unified Protocol or individually tailored) and type of support (by a specific therapist or by a team): (1) Unified Protocol with weekly support by a specific therapist, (2) Unified Protocol with weekly support by the team, (3) Individually tailored treatment with weekly support by a specific therapist, (4) Individually tailored treatment with weekly support by the team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Unified Protocol, support by a specific therapist (Experimental): The participants receive eight weeks of ICBT, based on the treatment manual Unified Protocol by David Barlow and colleagues (2013), with weekly support by a specific therapist that follow the individual participant through all treatment weeks. During the eight weeks, the participant will receive in total eight treatment modules.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy (ICBT)
- Unified Protocol, support by a team (Experimental): The participants receive eight weeks of ICBT, based on the treatment manual Unified Protocol by David Barlow and colleagues (2013), with weekly support by a team of therapists. This arm implies that the participant will get support from different therapists each week. During the eight weeks, the participant will receive in total eight treatment modules.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy (ICBT)
- Individually tailored treatment, support by a specific therapist (Experimental): The participants receive ICBT in an individually tailored format, where they get to select which modules they want to be included in their specific treatment. The participants are recommended to select eight modules (out of 25) and work with one modules each week, but this is only recommendations. In their treatment, weekly support by a specific therapist that follow the individual participant through all treatment weeks is included.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy (ICBT)
- Individually tailored treatment, support by team (Experimental): The participants receive ICBT in an individually tailored format, where they get to select which modules they want to be included in their specific treatment. The participants are recommended to select eight modules (out of 25) and work with one modules each week, but this is only recommendations. In their treatment, weekly support by a team of therapists is included. This arm implies that the participant will get support from different therapists each week.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy (ICBT)

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy (ICBT) — All participants get treatment and are thus included in experimental groups, no matter the randomization result. It consists of eight treatment weeks with weekly support. The treatment format will differ between the four groups, depending on type of treatment content and type of support.

SUMMARY:
The purpose of this study is to investigate the differences in treatment outcomes between individually tailored and transdiagnostic internet-based cognitive behavioral therapy (ICBT), as well as the differences between weekly support by a specific therapist and weekly support by a team. The target group is adults (18 years or older) who experience mild to moderate depression symptoms, anxiety, stress or other psychological symptoms. The ICBT, in both types of treatment contents, consists of modules that the participants will work with for eight weeks in total. Participants will be recruited in Sweden with nationwide recruitment.

DETAILED DESCRIPTION:
This study is a factorial randomized controlled trial with the aim to investigate ICBT with two kinds of treatment contents and two kinds of support. Participants will either be randomized to an individually tailored treatment, where they will be selecting their own modules that they wish to work with, or be randomized to a transdiagnostic treatment, that consists of Unified Protocol that is developed by David Barlow and colleagues. Participants will also be randomized to either get weekly support by one specific therapist or get support by "a team", meaning that the participant will get support from different therapists each week. In both kinds of support, the participant will have the opportunity to ask for support during the other times of the week as well.

Primary outcome measures are depression symptoms (measured with Beck Depression Inventory-II) and anxiety symptoms (measured with Beck Anxiety Inventory). Other, secondary, outcome measures used will for example be about stress symptoms, insomnia symptoms, and quality of life. Pre-treatment measurement, post-treatment measurement and one-year follow up is planned to be collected through an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Experience mild to moderate psychological symptoms or problems
* 18 years or older
* Ability to speak, read and write in Swedish
* Have access to the internet and a smartphone, computer or other device

Exclusion Criteria:

* Severe psychiatric or somatic illness that makes participation harder or impossible
* Ongoing addiction
* Acute suicidality
* Other ongoing psychological treatment
* Recent (within the latest month) changes in the dose of psychotropic medication or planned change of dose during the treatment weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Becks Depression Inventory-II | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of depressive symptoms. Range for the total sum is between 0 and 63 with a higher score indicating a higher level of depressive symptoms. Clinical ranges for minimal, mild, moderate and severe major depressive disorder are considered to be 0-13, 13-19, 20-28, and 29-63 points respectively.
Beck Anxiety Inventory | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of anxiety symptoms, consisting of 21 items. Range for the total sum is between 0 and 63, interpreted as minimal anxiety (0-7), mild anxiety (8-15), moderate anxiety (16-25) and severe anxiety (26-63).

SECONDARY OUTCOMES:
Perceived Stress Scale-14 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A questionnaire that aims to measure symptoms of stress. I contains 14 items that are scored on a range between 0 (never) to 4 (very often). The total score range is between 0-56 and a higher score reflects higher levels of perceived stress.
Insomnia Severity Index | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of insomnia severity and symptoms of disordered sleep. Norm score ranges include low likelihood of sleep problems (0 to 7 points), some sleep problems (8 to 14 points), moderate sleep problems (15 to 21 points), severe sleep problems (22 to 28 points).
Alcohol Use Disorder Identification Test | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. 10 items and scores ranging from 0-40 with higher scores indicating a higher level of alcohol use.
Brunnsviken Brief Quality of Life Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of quality of life with a total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.
Patient Health Questionnaire-15 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of somatic symptoms. It consists of 15 items for women and 14 items for men (because the item about "menstrual cramps or other problems with your periods" are removed). The symptoms are rated on a scale from 0 (not bothered) to 2 (bothered a lot). Total score ranges from 0 to 30 for women and 0 to 28 for men.
Goldberg's (1999) IPIP representation of Costa McCrae's (1992) NEO-PI-R Domains | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of neuroticism. It consists of 10 items, scored from 0 (Very inaccurate) to 4 (Very accurate).
InCharge Financial Distress/Financial Well-Being Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A measure aiming to measure distress related to the individual's economic situation. It contains of eight questions where the respondent gets to answer on a scale from 1 to 10. A higher score indicates lower economic distress.
Rosenberg's Self-esteem Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of self-esteem, consisting of ten items where five of them are positively and five of them are negatively worded. Sum scores range between 0-30. A higher score indicates higher self-esteem.

OTHER OUTCOMES:
Knowledge test (created by the research team) | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Knowledge test about cognitive behavior therapy and how strategies in cognitive behavior therapy can be applied in every day situations. It consists of 16 questions and the respondent gets three answer options while one of the alternatives are correct.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — University Hospital, Linkoeping
Locations (2):
- Sweden (2):
  - Linköping University, Linköping
  - Department of Behavioral Sciences and Learning, Linköping, Östergörland